CLINICAL TRIAL: NCT03521154
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, International Study of Osimertinib as Maintenance Therapy in Patients With Locally Advanced, Unresectable EGFR Mutation-positive Non-Small Cell Lung Cancer (Stage III) Whose Disease Has Not Progressed Following Definitive Platinum-based Chemoradiation Therapy (LAURA).
Brief Title: A Global Study to Assess the Effects of Osimertinib Following Chemoradiation in Patients With Stage III Unresectable Non-small Cell Lung Cancer (LAURA)
Acronym: LAURA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5160C00048; 2022-500860-36-00 (Registry Identifier: CTIS); 2018-001061-16 (EudraCT Number)
Record Dates: First submitted 2018-04-20; First posted 2018-05-11 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer (Stage III)
Keywords: Phase III; Osimertinib; Non Small Cell Lung Cancer (Stage III); Unresectable NSCLC; EGFR; chemoradiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osimertinib (Experimental): Osimertinib (80mg or 40mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Osimertinib 80mg/40mg
- Placebo Osimertinib (Placebo Comparator): Matching placebo for Osimertinib (80mg or 40mg orally, once daily), in accordance with the randomization schedule
  Interventions: Drug: Placebo Osimertinib 80mg/40mg

INTERVENTIONS:
Drug: Osimertinib 80mg/40mg — The initial dose of Osimertinib 80mg once daily can be reduced to 40mg once daily. Treatment can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Osimertinib
Drug: Placebo Osimertinib 80mg/40mg — The initial dose of Placebo Osimertinib 80mg once daily can be reduced to 40mg once daily.
  Treatment can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met
  Arms: Placebo Osimertinib

SUMMARY:
A global study to assess the efficacy and safety of osimertinib following chemoradiation in patients with stage III unresectable Epidermal Growth Factor Receptor Mutation Positive non-small cell lung cancer

DETAILED DESCRIPTION:
This is a phase 3 double-blind, randomized, placebo-controlled, study to assess the efficacy and safety of osimertinib following chemoradiation in patients with stage III unresectable EGFR mutation-positive NSCLC, including the most common EGFR sensitising mutations (Ex19Del and L858R), either alone or in combination with other EGFR mutations. Chemoradiation may have been given either given concurrently or sequentially. Patients whose disease has not progressed following chemoradiation will be randomised within 6 weeks of completion of chemoradiation to receive osimertinib or placebo in a 2:1 ratio, and treatment will be continued until disease progression, unacceptable toxicity or other discontinuation criteria are met. After progression, patients can be unblinded and may receive open-label osimertinib. After the final OS analysis, the study blind will be broken and patients still receiving open-label osimertinib will be supplied with open-label osimertinib by AstraZeneca for as long as their treating physician considers they are deriving clinical benefit.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged at least 18 years.
2. Patients with histologically documented NSCLC of predominantly non-squamous Pathology who present with locally advanced, unresectable (Stage III) disease (according to Version 8 of the International Association for the Study of Lung Cancer [IASLC] Staging Manual in Thoracic Oncology).
3. The tumor harbours one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations, assessed by cobas® EGFR Mutation Test v2 (Roche Diagnostics) or FoundationOne® test in a CLIA certified (USA sites) or an accredited local laboratory (sites outside of the USA) or by central testing (cobas® v2 only).
4. Patients must have received either concurrent chemoradiation or sequential chemoradiation including at least 2 cycles of platinum based chemotherapy and a total dose of radiation of 60 Gy ±10% (54 to 66 Gy).
5. Chemoradiation must be completed ≤6 weeks prior to randomization.
6. Patients must not have had disease progression during or following definitive platinum-based, chemoradiation therapy.
7. World Health Organization (WHO) performance status of 0 or 1.
8. Life expectancy >12 weeks at Day 1.
9. Female patients who are not abstinent (in line with the preferred and usual lifestyle choice) must be using adequate contraceptive measures, must not be breast feeding, and must have a negative pregnancy test prior to first dose of study drug; or female patients must have an evidence of non-childbearing potential.

Exclusion Criteria

1. Mixed small cell and non-small cell lung cancer histology
2. History of interstitial lung disease (ILD) prior to chemoradiation
3. Symptomatic pneumonitis following chemoradiation
4. Any unresolved toxicity Common Terminology Criteria for Adverse Events (CTCAE) > Grade 2 from the prior chemoradiation therapy
5. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
6. Inadequate bone marrow reserve or organ function
7. History of other malignancies, except: adequately treated non-melanoma skin cancer or lentigo maligna , curatively treated in-situ cancer, or other solid tumors curatively treated with no evidence of disease for > 5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
8. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib
10. Prior treatment with any prior chemotherapy, radiation therapy, immunotherapy or investigational agents for NSCLC outside of that received in the definitive setting for Stage III disease (chemotherapy and radiotherapy in SCRT and CCRT regimens is allowed for treatment of Stage III disease).
11. Prior treatment with EGFR-TKI therapy
12. Major surgery as defined by the investigator within 4 weeks of the first dose of study drug.
13. Patients currently receiving (unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 weeks prior to receiving the first dose of study drug).
14. Contraindication to MRI, including but not limited to, claustrophobia, pace makers, metal implants, intracranial surgical clips and metal foreign bodies

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2027-04-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh S Ramalingam, MD, Principal Investigator — Emory University School of Medicine, Atlanta, U.S.; Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital, Shanghai, China
Locations (91):
- United States (5):
  - Research Site, Duarte, California
  - Research Site, Atlanta, Georgia
  - Research Site, Florham Park, New Jersey
  - Research Site, Salt Lake City, Utah
  - Research Site, Madison, Wisconsin
- Argentina (4):
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- China (11):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Linhai
  - Research Site, Shanghai
  - Research Site, Ürümqi
  - Research Site, Wuhan
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Pécs
- India (7):
  - Research Site, Bangalore
  - Research Site, Gūrgaon
  - Research Site, Hubli
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Nashik
  - Research Site, New Delhi
- Japan (13):
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
- Research Site, Mérida, Mexico
- Peru (2):
  - Research Site, Lima
  - Research Site, San Isidro
- Russia (7):
  - Research Site, Kazan'
  - Research Site, Kostroma
  - Research Site, Moscow
  - Research Site, Novisibirsk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, San Sebastián
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Lampang
  - Research Site, Mueang
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Lu S, Kato T, Dong X, Ahn MJ, Quang LV, Soparattanapaisarn N, Inoue T, Wang CL, Huang M, Yang JC, Cobo M, Ozguroglu M, Casarini I, Khiem DV, Sriuranpong V, Cronemberger E, Takahashi T, Runglodvatana Y, Chen M, Huang X, Grainger E, Ghiorghiu D, van der Gronde T, Ramalingam SS; LAURA Trial Investigators. Osimertinib after Chemoradiotherapy in Stage III EGFR-Mutated NSCLC. N Engl J Med. 2024 Aug 15;391(7):585-597. doi: 10.1056/NEJMoa2402614. Epub 2024 Jun 2. PMID 38828946
- [Derived] Tu CY, Hsia TC, Lin YC, Liang JA, Li CC, Chien CR. Efficacy of Definitive Radiotherapy for Patients with Clinical Stage IIIB or IIIC Lung Adenocarcinoma and Epidermal Growth Factor Receptor (EGFR) Mutations Treated Using First- or Second-Generation EGFR Tyrosine Kinase Inhibitors. Can Respir J. 2024 Mar 5;2024:8889536. doi: 10.1155/2024/8889536. eCollection 2024. PMID 38476120
- [Derived] Lu S, Casarini I, Kato T, Cobo M, Ozguroglu M, Hodge R, van der Gronde T, Saggese M, Ramalingam SS. Osimertinib Maintenance After Definitive Chemoradiation in Patients With Unresectable EGFR Mutation Positive Stage III Non-small-cell Lung Cancer: LAURA Trial in Progress. Clin Lung Cancer. 2021 Jul;22(4):371-375. doi: 10.1016/j.cllc.2020.11.004. Epub 2021 Jan 6. PMID 33558193
- See also: D5160C00048_CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00048&attachmentIdentifier=d2981375-6416-4cae-bdc2-c103341ff3e6&fileName=D5160C00048_CSP_redacted.pdf&versionIdentifier=
- See also: D5160C00048_SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00048&attachmentIdentifier=4cc3eadf-3988-423d-9525-694fc3959131&fileName=D5160C00048_SAP_redacted.pdf&versionIdentifier=
- See also: D5160C00048_CSR synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00048&attachmentIdentifier=187ae97f-7617-494a-a48a-9326e63b829c&fileName=D5160C00048_CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients assigned to osimertinib may continue to receive osimertinib if, in the opinion of their treating physician, they are continuing to derive clinical benefit. Patients receiving placebo may receive open-label osimertinib, in accordance with local clinical practice and the judgement of their treating physician. For all patients, post-progression treatment with AZ-supply osimertinib may continue as long as the treating physician considers the patient to be deriving clinical benefit
Groups:
- Osimertinib: 80mg once daily tablet
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Osimertinib | Placebo
Started | 143 | 73
Completed | 32 | 21
Not Completed | 111 | 52
Not completed — Ongoing study at data cut-off | 111 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osimertinib | Placebo | Total
Number analyzed (Participants) | 143 | 73 | 216
Age, Continuous [Median (Full Range); unit: Years] | 62 [36 to 84] | 64 [37 to 83] | 62.5 [36 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 42 | 132
  Male | 53 | 31 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 13
  Not Hispanic or Latino | 132 | 71 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 116 | 62 | 178
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 10 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by Blinded Independent Central Review (BICR)
Description: Time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on BICR assessment according to RECIST v1.1
Time Frame: Every 8 weeks for first 48 weeks, then every 12 weeks until BICR-confirmed radiological disease progression. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | 39.13 [31.51 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of 95% confidence interval to be calculated | 5.55 [3.71 to 7.43]
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.10 to 0.24] — A hazard ratio < 1 favours osimertinib

2. Secondary Outcome: Number of Participants With Progression-free Survival (PFS) Events in Patients With EGFR Ex19del or L858R Mutation
Description: Number of PFS events (PFS is time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on BICR assessment according to RECIST v1.1)
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Participants
  Ex19Del positive: number analyzed (Participants) | 74 | 43
  Ex19Del positive | 26 | 39
  L858R positive: number analyzed (Participants) | 68 | 30
  L858R positive | 31 | 24
  Missing: number analyzed (Participants) | 1 | 0
  Missing | 0 | 0
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; PFS in Ex19Del positive patients; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.10 to 0.29] — A hazard ratio < 1 favours osimertinib
Statistical Analysis 2: Comparison: Osimertinib vs Placebo; PFS in L858R positive patients; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.32, 95% CI [0.19 to 0.56] — A hazard ratio < 1 favours osimertinib

3. Secondary Outcome: Number of Participants With Progression-free Survival (PFS) Events in Patients With EGFR Mutations Ex19del or L858R Detectable in Plasma-derived ctDNA
Description: Number of PFS events (PFS is time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on blinded independent central review (BICR) assessment according to RECIST v1.1)
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Participants
  EGFR mutation-positive: number analyzed (Participants) | 10 | 4
  EGFR mutation-positive | 4 | 4
  EGFR mutation-negative: number analyzed (Participants) | 113 | 58
  EGFR mutation-negative | 42 | 51
  EGFR mutation-unknown: number analyzed (Participants) | 20 | 11
  EGFR mutation-unknown | 11 | 8
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Negative at screening; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.15 to 0.34] — A hazard ratio < 1 favours osimertinib

4. Secondary Outcome: Central Nervous System (CNS) Progression-free Survival (PFS) by Blinded Independent Central Review (BICR)
Description: Time from randomisation until the date of CNS disease progression or death (by any cause in the absence of CNS progression) regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on CNS BICR assessment according to RECIST v1.1
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | NA [NA to NA] — NA - Not calculated as insufficient number of events to enable the median and 95% confidence interval to be calculated | 14.88 [7.36 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of the 95% confidence interval to be calculated
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.09 to 0.32] — A hazard ratio < 1 favours osimertinib

5. Secondary Outcome: Overall Survival (Count)
Description: Number of patients with Overall Survival (OS), the time from the date of randomisation until date of death by any cause
Time Frame: Date of randomisation to date of death by any cause. Assessed up to a maximum of approximately 63 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Participants
  Died | 28 | 15
  Censored (includes participants still in survival follow up and terminated prior to death) | 115 | 58

6. Secondary Outcome: Overall Survival (Duration)
Description: Time from the date of randomisation until death by any cause
Time Frame: Date of randomisation to date of death by any cause. Assessed up to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | 53.95 [46.49 to NA] — NA - Not calculated as insufficient number of events to enable upper limit of 95% confidence interval to be calculated | NA [42.05 to NA] — NA - Not calculated as insufficient number of events to enable median and upper limit of 95% confidence interval to be calculated
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p = 0.530, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.42 to 1.56] — A hazard ratio < 1 favours osimertinib

7. Secondary Outcome: Objective Response Rate by Blinded Independent Central Review (BICR)
Description: Percentage of evaluable patients with at least one BICR assessed visit response of complete response (CR) or partial response (PR). CR defined as disappearance of all target lesions (TL) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm. PR defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline sum of diameters). Responses include both confirmed and unconfirmed BICR responses
Time Frame: Every 8 weeks for first 48 weeks, then every 12 weeks until radiological disease progression. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
% of participants | 57.3 [48.8 to 65.6] | 32.9 [22.3 to 44.9]
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.54 to 5.08] — An odds ratio > 1 favours osimertinib

8. Secondary Outcome: Duration of Response, Unconfirmed by Blinded Independent Central Review (BICR)
Description: Date of PFS event - date of first unconfirmed response + 1 day (and expressed in months) for unconfirmed responses only
Time Frame: as for outcome 7
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 82 | 24
Months | 36.9 [17.9 to NA] — NA - Not calculated as insufficient number of events to enable 75% percentile to be calculated | 6.5 [3.2 to 9.0]

9. Secondary Outcome: Disease Control Rate by Blinded Independent Central Review (BICR)
Description: Percentage of patients who have a best overall response of complete response (CR), partial response (PR) or stable disease (SD) as assessed by BICR
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
% of participants | 88.8 [82.5 to 93.5] | 79.5 [68.4 to 88.0]
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p = 0.069, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.94 to 4.47] — An odds ratio > 1 favours osimertinib

10. Secondary Outcome: Tumour Shrinkage by Blinded Independent Central Review (BICR)
Description: Depth of response (or tumour shrinkage or change in tumour size) was assessed using BICR responses in target lesions. The best change in tumour size is the largest decrease from baseline or the smallest increase from baseline in the absence of a reduction
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Full Range); unit: % change from baseline
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 133 | 70
% change from baseline | -43.3 [-100 to 144] | -21.9 [-100 to 23]

11. Secondary Outcome: Proportion With Tumour Shrinkage by Blinded Independent Central Review (BICR)
Description: Proportion with depth of response (or tumour shrinkage or change in tumour size)
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: Proportion of participants
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Proportion of participants
  Proportion with reduction | 0.92 | 0.83
  Proportion with reduction > 30% | 0.65 | 0.40
  Proportion with reduction > 50% | 0.43 | 0.11
  Proportion with reduction > 75% | 0.18 | 0.09

12. Secondary Outcome: Time to Death or Distant Metastases by Blinded Independent Central Review (BICR)
Description: Time from the date of randomisation until the first date of distant metastases or date of death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that is detected on a scan that is anywhere other than lung or regional lymph node according to RECIST v1.1 or proven by biopsy
Time Frame: Time from randomisation to the date of distant metastases or death. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | NA [39.29 to NA] — NA - Not calculated as median not reached and insufficient number of events to enable upper limit of 95% confidence interval to be calculated | 13.04 [9.03 to NA] — NA - Not calculated as insufficient number of events to enable upper limit of 95% confidence interval to be calculated
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.11 to 0.38] — A hazard ratio < 1 favours osimertinib

13. Secondary Outcome: Time to Study Treatment Discontinuation
Description: Time from randomisation to the earlier of the date of study treatment discontinuation (regardless of the reason for study treatment discontinuation) or death (i.e. date of study treatment discontinuation/death or censoring - date of randomisation + 1 day, expressed in months)
Time Frame: Time from randomisation to the earlier of the date of study treatment discontinuation or death. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | 40.28 [32.72 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of the 95% confidence interval to be calculated | 8.31 [6.14 to 11.10]
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.14 to 0.32] — A hazard ratio < 1 favours osimertinib

14. Secondary Outcome: Time to First Subsequent Treatment
Description: Time from the date of randomisation to the earlier of the date of anti-cancer therapy start date following study drug discontinuation or death
Time Frame: Time from randomisation to the start of first subsequent anti-cancer therapy or death. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | 43.83 [38.87 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of 95% confidence interval to be calculated | 9.46 [6.60 to 11.53]
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.08 to 0.21] — A hazard ratio < 1 favours osimertinib

15. Secondary Outcome: Time to Second Subsequent Treatment
Description: Time from the date of randomisation to the earlier of the second subsequent anti-cancer therapy start date following study drug discontinuation or death
Time Frame: Time from randomisation to the start of second subsequent anti-cancer therapy or death. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | NA [44.42 to NA] — NA - Not calculated as insufficient number of events to enable the median and upper limit of 95% confidence interval to be calculated | 47.38 [34.14 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of 95% confidence interval to be calculated
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p = 0.022, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.28 to 0.91] — A hazard ratio < 1 favours osimertinib

16. Secondary Outcome: Second Progression-free Survival (PFS2)
Description: Time from randomisation to the earliest progression event following first objective disease progression, subsequent to the first subsequent therapy, or death.
Time Frame: Every 8 weeks for first 48 weeks, then every 12 weeks. Assessed up to date of DCO (05Jan24) to a maximum of approximately 63 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib | Placebo
Number analyzed (Participants) | 143 | 73
Months | 48.20 [44.42 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of 95% confidence interval to be calculated | 47.38 [28.22 to NA] — NA - Not calculated as insufficient number of events to enable the upper limit of 95% confidence interval to be calculated
Statistical Analysis 1: Comparison: Osimertinib vs Placebo; Test type: Superiority; p = 0.088, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.35 to 1.08] — A hazard ratio < 1 favours osimertinib

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent throughout the treatment period (maximum actual duration of 62.4 and 56.2 months for Osimertinib and Placebo respectively) up to and including 28 day follow up following last dose of study drug.
Description: The initial dose of osimertinib/placebo 80 mg QD could be reduced to 40 mg QD to allow for management of study treatment-related toxicities. Once the dose of osimertinib/placebo was reduced to 40 mg QD, the patient was to remain on the reduced dose until termination from study treatment
Arm/Group | Osimertinib | Placebo
All-Cause Mortality (participants affected / at risk) | 28/143 | 15/73
Serious Adverse Events (participants affected / at risk) | 55/143 | 11/73
Other Adverse Events (participants affected / at risk) | 129/143 | 54/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib (N=143) | Placebo (N=73)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis b (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 15 (15) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib (N=143) | Placebo (N=73)
Stomatitis (Gastrointestinal disorders) | 17 (20) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 13 (16) | 3 (3)
Covid-19 (Infections and infestations) | 28 (28) | 6 (6)
Herpes zoster (Infections and infestations) | 13 (13) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (9) | 0 (0)
Paronychia (Infections and infestations) | 24 (29) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 10 (18) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (13) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 55 (55) | 26 (27)
Alanine aminotransferase increased (Investigations) | 10 (12) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 8 (11) | 1 (1)
Platelet count decreased (Investigations) | 8 (14) | 0 (0)
White blood cell count decreased (Investigations) | 17 (35) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 21 (23) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (7)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (22) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (20) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 34 (40) | 10 (11)
Sinus tachycardia (Cardiac disorders) | 8 (12) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 51 (67) | 10 (11)

LIMITATIONS AND CAVEATS:
As per CSP Section 7.2, patient monitoring during treatment with open-label osimertinib is monitored by the investigator per local clinical guidance. Serious AEs and AESIs are reported in the eCRF but were not analyzed/tabulated at the time of primary analysis. Safety assessments are to be performed as per local clinical practice and not collected as part of study data capture in line with the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03521154/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03521154/SAP_001.pdf